CLINICAL TRIAL: NCT00559715
Title: Prevention of Vision Loss in Patients With Age-Related Neovascular Macular Degeneration by Intravitreal Injection of Bevacizumab and Ranibizumab in a Typical Outpatient Setting
Brief Title: Prevention of Vision Loss in Patients With Age-Related Macular Degeneration (AMD) by Intravitreal Injection of Bevacizumab and Ranibizumab
Acronym: VIBERA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum Bremen-Mitte, gGmbH (Other)
Collaborators: Kompetenzzentrum für Klinische Studien, Bremen (Unknown)
Responsible Party: Bernd Muehlbauer, Professor MD, Klinikum Bremen Mitte gGmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIBERA_2007-004721-23
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Age-Related Neovascular Macular Degeneration
Keywords: bevacizumab; ranibizumab; macular degeneration; age-related; neovascular; intravitreal injection; vision loss; outpatient setting
MeSH Terms: conditions — Macular Degeneration; Vision Disorders | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: bevacizumab
- B (Active Comparator)
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: bevacizumab — 1.25 mg intravitreally monthly/on demand
  Other Names: Avastin®
  Arms: A
Drug: ranibizumab — 0.5 mg intravitreally monthly/on demand
  Other Names: Lucentis®
  Arms: B

SUMMARY:
The study is designed to demonstrate the therapeutic non-inferiority of the recombinant humanized monoclonal VEGF antibody bevacizumab administered by intravitreal injection in the treatment of AMD in comparison to the related fragment ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients with visual impairment (best corrected visual acuity of 20/40 to 20/320 (Snellen equivalent, ETDRS chart)) due to an active primary or recurrent CNV associated with age-related macular degeneration involving the foveal center, presenting with either:

  * a classical / predominantly classical lesion with largest diameter of SNVM smaller than greatest distance between major temporal vascular arcades or
  * a minimally classical lesion or an occult lesion with no classic choroidal neovascularization

Exclusion Criteria:

* Known or suspected hypersensitivity to ranibizumab or bevacizumab
* Participation in any clinical trial within the last 4 weeks
* Previous participation in a clinical trial (for either eye) involving antiangiogenic drugs (pegaptanib, bevacizumab ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Previous laser photocoagulation (juxtafoveal or extrafoveal) in the study eye
* History of vitreoretinal surgery in the study eye
* History of submacular surgery or other surgical intervention for AMD in the study eye
* Subretinal hemorrhage in the study eye that involves the fovea, if the size of the hemorrhage is either 50% or more of the total lesion area or 1 or more disc areas in size
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either:
* require medical or surgical intervention during the 24-month study period to prevent or treat visual loss that might result from that condition, or
* if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 24-month study period
* Active intraocular, ocular, or periocular inflammation (any grade "trace" or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure [IOP] of 30 mmHg or more despite treatment with antiglaucoma medications)
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* History of allergy to fluorescein, not amenable to treatment with diphenhydramine
* Inability to obtain fundus photographs or FA of sufficient quality to be analyzed and graded by the blinded evaluation center
* Inability to comply with study or follow-up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a loss of fewer than 15 letters at month 12 | 1 year

SECONDARY OUTCOMES:
Proportion of patients with a loss of fewer than 15 letters at month 24 | 2 years
Mean change from baseline in BCVA at month 12 (IA) and month 24 | 2 years
Proportion of patients with a treatment-free interval of at least 3 months' duration at any time point following month 2 | 2 years
Number of doses of the study drugs | 2 years
Drop out rates | 2 years
Rate of non-responders | 2 years
Retinal lesions | 2 years
Adverse Events | 2 years
Quality of Life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Muehlbauer, Professor MD, Principal Investigator — Department of Pharmacology, Klinikum Bremen Mitte, Bremen, Germany
Locations (1):
- Department of Pharmacology at Klinikum Bremen Mitte, Bremen, Germany